CLINICAL TRIAL: NCT02084056
Title: Bioequivalence of a Fixed Dose Combination Tablet of Linagliptin/Metformin Extended Release (2.5 mg/1000 mg) Compared With the Free Combination of Linagliptin and Metformin Extended Release Tablets in Healthy Subjects (an Open-label, Randomised, Single Dose, Two-way Crossover Trial)
Brief Title: Bioequivalence of a FDC Tablet of Linagliptin/Metformin (2.5mg/1000mg) Extended Release in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1288.11; 2013-005144-28 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Results first posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin; Metformin

ARMS (4):
- FDC first, fasted (Experimental): Linagliptin/Metformin FDC followed by single tablets of linagliptin and metformin, fasted
  Interventions: Drug: Linagliptin; Drug: Metformin; Drug: Linagliptin/Metformin FDC
- Single tablets first, fasted (Experimental): single tablets of linagliptin and metformin followed by Linagliptin/Metformin FDC, fasted
  Interventions: Drug: Linagliptin; Drug: Metformin; Drug: Linagliptin/Metformin FDC
- FDC first, fed (Experimental): Linagliptin/Metformin FDC followed by single tablets of linagliptin and metformin, fed
  Interventions: Drug: Linagliptin; Drug: Metformin; Drug: Linagliptin/Metformin FDC
- Single tablets first, fed (Experimental): single tablets of linagliptin and metformin followed by Linagliptin/Metformin FDC, fed
  Interventions: Drug: Linagliptin; Drug: Metformin; Drug: Linagliptin/Metformin FDC

INTERVENTIONS:
Drug: Linagliptin — Linagliptin
Drug: Metformin — Metformin
Drug: Linagliptin/Metformin FDC — Linagliptin/Metformin FDC

SUMMARY:
The purpose of this trial is to demonstrate bioequivalence of a newly developed fixed dose combination (FDC) tablet containing linagliptin and metformin extended release compared to the free combination of linagliptin and metformin extended release.

ELIGIBILITY:
Inclusion criteria:

- Healthy male or female subjects

Exclusion criteria:

- Any relevant deviation from healthy condition

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1288.11.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in two parts. Part 1: Fasting study Part 2: Fed Study
Groups:
- FDC 2000 Fasted / L+M 2000 Fasted: Linagliptin+ Metformin Fixed dose combination (FDC)-(T fasted): 2X2.5 mg linagliptin/1000 mg metformin Extended Release (XR) (given as FDC tablet) followed by 5 mg linagliptin and 2000 mg metformin XR (given as 1 tablet 5 mg linagliptin and 4 tablets 500 mg metformin XR; R fasted) orally with 240 mL of water after an overnight fast of at least 10 h.
  Where, L+M = Linagliptin 5mg+Metformin XR 2000mg
- L+M 2000 Fasted / FDC 2000 Fasted: Linagliptin+ Metformin-(R fasted): 5 mg linagliptin and 2000 mg metformin XR (given as 1 tablet 5 mg linagliptin and 4 tablets 500 mg metformin XR) followed by Linagliptin+ Metformin (FDC)-(T fasted): 2X2.5 mg linagliptin/1000 mg metformin XR orally with 240 mL of water after an overnight fast of at least 10 h.
  Where, L+M = Linagliptin 5mg+Metformin XR 2000mg
- FDC 2000 Fed / L+M 2000 Fed: Linagliptin+ Metformin (FDC)-(T fed): 2X2.5 mg linagliptin/1000 mg metformin XR (given as FDC tablet) followed by 5 mg linagliptin and 2000 mg metformin XR (given as 1 tablet 5 mg linagliptin and 4 tablets 500 mg metformin XR; R fed) orally with 240 mL of water after after a high-fat, high-calorie meal.
  Where, L+M = Linagliptin 5mg+Metformin XR 2000mg
- L+M 2000 Fed / FDC 2000 Fed: Linagliptin+ Metformin-(R fed): 5 mg linagliptin and 2000 mg metformin XR (given as 1 tablet 5 mg linagliptin and 4 tablets 500 mg metformin XR) followed by Linagliptin+ Metformin (FDC)-(T fed): 2X2.5 mg linagliptin/1000 mg metformin XR orally with 240 mL of water after a high-fat, high-calorie meal.
  Where, L+M = Linagliptin 5mg+Metformin XR 2000mg
Period: Treatment Period 1 (4 Days)
Arm/Group | FDC 2000 Fasted / L+M 2000 Fasted | L+M 2000 Fasted / FDC 2000 Fasted | FDC 2000 Fed / L+M 2000 Fed | L+M 2000 Fed / FDC 2000 Fed
Started | 28 | 30 | 8 | 8
Completed | 27 | 30 | 8 | 8
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Washout Period 1 (35 Days)
Arm/Group | FDC 2000 Fasted / L+M 2000 Fasted | L+M 2000 Fasted / FDC 2000 Fasted | FDC 2000 Fed / L+M 2000 Fed | L+M 2000 Fed / FDC 2000 Fed
Started | 27 | 30 | 8 | 8
Completed | 26 | 30 | 8 | 8
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Treatment Period 2 (4 Days)
Arm/Group | FDC 2000 Fasted / L+M 2000 Fasted | L+M 2000 Fasted / FDC 2000 Fasted | FDC 2000 Fed / L+M 2000 Fed | L+M 2000 Fed / FDC 2000 Fed
Started | 26 | 30 | 8 | 8
Completed | 26 | 30 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set: All randomised subjects who received 1 dose of trial medication were included in the treated set.
Groups:
- FDC 2000 Fasted or L+M 2000 Fasted: The subjects in Part 1 were randomly allocated to 1 of the 2 treatment sequences T fasted_R fasted or R fasted_T fasted.
  FDC 2000 fasted (T fasted): 2X2.5 mg linagliptin/1000 mg metformin XR (given as FDC tablet) orally with 240 mL of water after an overnight fast of at least 10 h.
  L+M 2000 fasted (R fasted): 5 mg linagliptin and 2000 mg metformin XR (given as 1 tablet 5 mg linagliptin and 4 tablets 500 mg metformin XR; R fasted) orally with 240 mL of water after an overnight fast of at least 10 h.
  Where, L+M = Linagliptin 5mg+Metformin XR 2000mg
- FDC 2000 Fed or L+M 2000 Fed: The subjects in Part 2 were randomly allocated to 1 of the 2 treatment sequences T fed_R fed or R fed_T fed.
  FDC 2000 fed (T fed): 2X2.5 mg linagliptin/1000 mg metformin XR (given as FDC tablet) orally with 240 mL of water after a high-fat, high-calorie meal.
  L+M 2000 fed (R fed): 5 mg linagliptin and 2000 mg metformin XR (given as 1 tablet 5 mg linagliptin and 4 tablets 500 mg metformin XR; R fed) orally with 240 mL of water after a high-fat, high-calorie meal.
  Where, L+M = Linagliptin 5mg+Metformin XR 2000mg
- Total: Total of all reporting groups
Arm/Group | FDC 2000 Fasted or L+M 2000 Fasted | FDC 2000 Fed or L+M 2000 Fed | Total
Number analyzed (Participants) | 58 | 16 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (9.8) | 32.6 (8.2) | 33.0 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 7 | 45
  Male | 20 | 9 | 29

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Linagliptin in Plasma Over the Time Interval From 0 to 72 Hours (AUC0-72)
Description: AUC 0-72 (area under the concentration-time curve of Linagliptin in plasma from 0 to 72 hours) The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: 1 hour (h) before drug administration and 20 minutes (min), 40min, 1h,1h 30min, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h,34h, 48h and 72h after drug administration
Population: PKS2000 Fast and PKS2000 Fed, consists of the subjects who provided at least 1 observation for at least 1 primary endpoint without Important protocol violations with respect to the statistical evaluation of pharmacokinetic endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- L+M 2000 Fasted: 5 mg linagliptin/2000 mg metformin XR (given as 1 tablet 5 mg linagliptin and 4 tablets 500 mg metformin XR; R fasted) orally with 240 mL of water after an overnight fast of at least 10 h.
- FDC 2000 Fasted: 5 mg linagliptin and 2000 mg metformin XR FDC (given as 2 tablet 2.5 mg linagliptin and 1000 mg metformin XR) orally with 240 mL of water after an overnight fast of at least 10 h.
- L+M 2000 Fed: 5 mg linagliptin/2000 mg metformin XR given as 1 tablet 5 mg linagliptin and 4 tablets 500 mg metformin XR; R fed) orally with 240 mL of water after a high-fat, high-calorie meal.
- FDC 2000 Fed: 5 mg linagliptin and 2000 mg metformin XR FDC (given as 2 tablet 2.5 mg linagliptin and 1000 mg metformin XR) orally with 240 mL of water after a high-fat, high-calorie meal.
Arm/Group | L+M 2000 Fasted | FDC 2000 Fasted | L+M 2000 Fed | FDC 2000 Fed
Number analyzed (Participants) | 55 | 57 | 16 | 15
nmol*h/L | 278.460 (9.1) | 288.709 (9.1) | 264.509 (12.7) | 268.814 (12.7)
Statistical Analysis 1: Comparison: L+M 2000 Fasted vs FDC 2000 Fasted; Test type: Non-Inferiority or Equivalence — The assessment of bioequivalence was based upon 2-sided 90% confidence intervals (CIs) for the ratios of the geometric means (FDC/free combination) using an acceptance range of 80.00 to 125.00%; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 103.68, 90% CI 2-sided [100.703 to 106.747], Standard Error of Mean 1.018 — Ratio of (FDC 2000 fasted/ L+M 2000 fasted)
Statistical Analysis 2: Comparison: L+M 2000 Fed vs FDC 2000 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0003, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 101.63, 90% CI 2-sided [93.721 to 110.202], Standard Error of Mean 1.047 — Ratio of (FDC 2000 fed/ L+M 2000 fed)

2. Primary Outcome: Maximum Measured Concentration of Linagliptin in Plasma (Cmax)
Description: Cmax (maximum measured concentration of Linagliptin in plasma) The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | L+M 2000 Fasted | FDC 2000 Fasted | L+M 2000 Fed | FDC 2000 Fed
Number analyzed (Participants) | 55 | 57 | 16 | 15
nmol/L | 8.274 (19.6) | 9.480 (19.6) | 6.729 (20.1) | 6.613 (20.1)
Statistical Analysis 1: Comparison: L+M 2000 Fasted vs FDC 2000 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0113, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 114.58, 90% CI 2-sided [107.687 to 121.908], Standard Error of Mean 1.038 — Ratio of (FDC 2000 fasted/ L+M 2000 fasted)
Statistical Analysis 2: Comparison: L+M 2000 Fed vs FDC 2000 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0064, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 98.28, 90% CI 2-sided [86.543 to 111.609], Standard Error of Mean 1.075 — Ratio of (FDC 2000 fed/ L+M 2000 fed)

3. Primary Outcome: Area Under the Concentration-time Curve of Metformin in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: AUC 0-tz (Area under the concentration-time curve of metformin in plasma over the time interval from 0 to the last quantifiable data point) The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | L+M 2000 Fasted | FDC 2000 Fasted | L+M 2000 Fed | FDC 2000 Fed
Number analyzed (Participants) | 56 | 56 | 15 | 15
ng*h/mL | 12028.27 (17.6) | 11601.19 (17.6) | 20411.01 (11.7) | 19952.61 (11.7)
Statistical Analysis 1: Comparison: L+M 2000 Fasted vs FDC 2000 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 96.45, 90% CI 2-sided [91.23 to 101.97], Standard Error of Mean 1.03 — Ratio of (FDC 2000 fasted/ L+M 2000 fasted)
Statistical Analysis 2: Comparison: L+M 2000 Fed vs FDC 2000 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0002, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 97.75, 90% CI 2-sided [90.47 to 105.63], Standard Error of Mean 1.04 — Ratio of (FDC 2000 fed/ L+M 2000 fed)

4. Primary Outcome: Cmax of Metformin in Plasma
Description: Cmax (maximum measured concentration of Metformin in plasma) The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | L+M 2000 Fasted | FDC 2000 Fasted | L+M 2000 Fed | FDC 2000 Fed
Number analyzed (Participants) | 56 | 57 | 15 | 15
ng/mL | 1516.558 (19.9) | 1485.642 (19.9) | 1571.040 (13.8) | 1662.954 (13.8)
Statistical Analysis 1: Comparison: L+M 2000 Fasted vs FDC 2000 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 97.96, 90% CI 2-sided [92.046 to 104.257], Standard Error of Mean 1.038 — Ratio of (FDC 2000 fasted/ L+M 2000 fasted)
Statistical Analysis 2: Comparison: L+M 2000 Fed vs FDC 2000 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0030, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 105.85, 90% CI 2-sided [96.705 to 115.861], Standard Error of Mean 1.053 — Ratio of (FDC 2000 fed/ L+M 2000 fed)

5. Secondary Outcome: Area Under the Concentration-time Curve of Linagliptin in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-inf)
Description: AUC0-inf (area under the concentration-time curve of linagliptin in plasma over the time interval from 0 extrapolated to infinity) for Linagliptin.
  The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | L+M 2000 Fasted | FDC 2000 Fasted | L+M 2000 Fed | FDC 2000 Fed
Number analyzed (Participants) | 55 | 57 | 16 | 15
nmol*h/L | 457.780 (15.8) | 473.704 (15.8) | 445.884 (16.7) | 451.888 (16.7)
Statistical Analysis 1: Comparison: L+M 2000 Fasted vs FDC 2000 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 103.48, 90% CI 2-sided [98.426 to 108.790], Standard Error of Mean 1.030 — Ratio of (FDC 2000 fasted/ L+M 2000 fasted)
Statistical Analysis 2: Comparison: L+M 2000 Fed vs FDC 2000 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0019, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 101.35, 90% CI 2-sided [91.130 to 112.708], Standard Error of Mean 1.062 — Ratio of (FDC 2000 fed/ L+M 2000 fed)

6. Secondary Outcome: AUC0-inf of Metformin in Plasma
Description: AUC0-inf(area under the concentration-time curve of the metformin in plasma over the time interval from 0 extrapolated to infinity) for Metformin.
  The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: as for outcome 1
Population: PKS 2000 fast and PKS 2000 fed, included all treated subjects in Part 1 and Part 2, respectively, who provided at least 1 observation for at least 1 primary endpoint, without important protocol violations regarding the statistical evaluation of pharmacokinetic endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | L+M 2000 Fasted | FDC 2000 Fasted | L+M 2000 Fed | FDC 2000 Fed
Number analyzed (Participants) | 56 | 56 | 15 | 15
ng*h/mL | 12736.87 (19.7) | 12162.37 (19.7) | 20721.20 (11.9) | 20346.34 (11.9)
Statistical Analysis 1: Comparison: L+M 2000 Fasted vs FDC 2000 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 95.49, 90% CI 2-sided [89.73 to 101.62], Standard Error of Mean 1.04 — Ratio of (FDC 2000 fasted/ L+M 2000 fasted)
Statistical Analysis 2: Comparison: L+M 2000 Fed vs FDC 2000 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0002, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 98.19, 90% CI 2-sided [90.73 to 106.27], Standard Error of Mean 1.05 — Ratio of (FDC 2000 fed/ L+M 2000 fed)

ADVERSE EVENTS:
Time Frame: From the first drug administration for at least 7 days after the last drug administration, up to 47 days.
Arm/Group | L+M 2000 Fasted | FDC 2000 Fasted | L+M 2000 Fed | FDC 2000 Fed
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/58 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 20/56 | 24/58 | 8/16 | 5/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | L+M 2000 Fasted (N=56) | FDC 2000 Fasted (N=58) | L+M 2000 Fed (N=16) | FDC 2000 Fed (N=16)
Abdominal pain (Gastrointestinal disorders) | 3 | 6 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 4 | 1
Nausea (Gastrointestinal disorders) | 2 | 5 | 2 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Discomfort (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 0 | 0
Headache (Nervous system disorders) | 11 | 9 | 3 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes